CLINICAL TRIAL: NCT04861246
Title: Evaluation of Laser Treatment for Benign Pigmented Lesions by Non-invasive, Cellular Resolution Optical Coherence Tomography
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow recruitment due to covid-19 disruptions
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Collaborators: Apollo Medical Optics, Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2020-08-006C
Record Dates: First submitted 2021-04-26; First posted 2021-04-27 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Benign Pigmented Lesions
Keywords: Optical Coherence Tomograohy; Non-invasive image system; Cellular level resolution; Full-Field OCT; Hyperpigmentation
MeSH Terms: conditions — Hyperpigmentation | interventions — Lasers

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Epidermal pigmented lesion
  Interventions: Device: Laser; Device: ApolloVue® S100 Image System; Device: VISIA®

INTERVENTIONS:
Device: Laser — The device will be used to do Laser treatment. To compare the therapeutic effect to laser treatment before and post treatment for 14 and 60 days.
Device: ApolloVue® S100 Image System — The device is an in vivo non-invasive optical coherence tomography and will be used to obtain OCT images before and after laser treatment of skin.
Device: VISIA® — The device is skin analysis system and will be used to obtain before and after images of laser treatment.

SUMMARY:
In recent years, with the maturity of laser technology, laser therapy is one of the popular options for the treatment of pigment diseases. The absorption spectrum of melanin ranges from 300 to 1,000 nm. In past studies, the 532 nm Q-switched Nd:YAG laser is effective for the treatment of superficial melanin. But there are still some side effects in laser treatment, such as post-inflammation pigmentation (PIH), depigmentation, skin redness, etc., and PIH is particularly likely to occur on darker skin. However, there is still no good evidence as to what factors or laser treatments can cause PIH.

Therefore, in this study, we will use ApolloVue® S100 Image System (ApolloVue® S100 Image System is a medical device class II) to scan before and after skin of laser treatment to observe the changes in the skin condition. By observing and analyzing these changes, as a evaluation of predictors or prognostic factors after laser treatment and whether PIH will occur.

ELIGIBILITY:
Inclusion Criteria:

* Age ≧ 20
* Both gender are accepted
* Subject with pigmented diseases
* The pigmented lesions which participating the trial were not treated in the last 12 months
* Accepts not to expose the face to sunlight or artificial UV rays during the study
* Is willing to comply with all requirements of the study including being photographed, following post treatment care and attending all treatment and follow up visits
* During the trial period, willing to use the maintenance and sunscreen products provided in this trial for care

Exclusion Criteria:

* Pregnant woman or woman wishing to be pregnant during the study, or during breastfeeding period
* Has any condition which, in the investigator's opinion, would make it unsafe for participating in this research study
* Has systemic skin disorders or infections
* Is enrolled or accepted other investigational drug or medical device

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2022-03-22 (Actual); Study Completion 2022-03-22 (Actual)

PRIMARY OUTCOMES:
Static Physician's Global Assessment (PGA) | one and a half years
  Static PGA is often used to evaluate disease severity of psoriasis. In recent years, this evaluation index has also been applied to pigmented diseases, such as solar lentigo, melasma, and vitiligo. In this trial, Static PGA divides the severity of pigmented diseases into 0~8.
  1. 0: Extremely lighter than pigment of surrounding skin (completely depigmented)
  2. 1: markedly lighter than pigment of surrounding skin
  3. 2: moderately lighter than pigment of surrounding skin
  4. 3: slightly lighter than pigment of surrounding skin
  5. 4: equal with pigment of surrounding skin
  6. 5: slightly darker than pigment of surrounding skin
  7. 6: moderately darker than pigment of surrounding skin
  8. 7: markedly darker than pigment of surrounding skin
  9. 8: extremely darker than pigment of surrounding skin
Dynamic Physician's Global Assessment (PGA) | one and a half years
  Dynamic PGA is often used to evaluate the degree of improvement after treatment of the disease. In this trial, Dynamic PGA evaluates the degree of improvement after comparing with the state before treatment (baseline). The degree of improvement is divided into 0~5.
  1. 0: completely cleared of undesired pigment; no evidence of cosmetic deficit remaining; 100% improvement
  2. 1: significant clearance of undesired pigment; slight evidence of cosmetic deficit remaining; about 75% improvement
  3. 2: moderate clearance of undesired pigment; moderate evidence of cosmetic deficit remaining; about 50% improvement
  4. 3: slight clearance of undesired pigment; marked evidence of cosmetic deficit remaining; about 25% improvement
  5. 4: no change in cosmetic appearance from baseline
  6. 5: cosmetic appearance worse than at baseline
Subject satisfaction | one and a half years
  During the two follow-up visits after treatment, subjects will evaluate their satisfaction after treatment. In this trial, this evaluation form will be divided into 0 to 5 points according to the degree of improvement.
  1. 0: completely cleared of undesired pigment; no evidence of cosmetic deficit remaining; 100% improvement
  2. 1: significant clearance of undesired pigment; slight evidence of cosmetic deficit remaining; about 75% improvement
  3. 2: moderate clearance of undesired pigment; moderate evidence of cosmetic deficit remaining; about 50% improvement
  4. 3: slight clearance of undesired pigment; marked evidence of cosmetic deficit remaining; about 25% improvement
  5. 4: no change in cosmetic appearance from baseline
  6. 5: cosmetic appearance worse than at baseline

CONTACTS AND LOCATIONS:
Overall Officials: Cheng-Yuan Li, M.D., Principal Investigator — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Taipei Veterans General Hospital, Taipei, Beitou District, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vashi NA, Kundu RV. Facial hyperpigmentation: causes and treatment. Br J Dermatol. 2013 Oct;169 Suppl 3:41-56. doi: 10.1111/bjd.12536. PMID 24098900
- [Background] Vachiramon V, Panmanee W, Techapichetvanich T, Chanprapaph K. Comparison of Q-switched Nd: YAG laser and fractional carbon dioxide laser for the treatment of solar lentigines in Asians. Lasers Surg Med. 2016 Apr;48(4):354-9. doi: 10.1002/lsm.22472. Epub 2016 Jan 12. PMID 27096729
- [Background] Wang CC, Sue YM, Yang CH, Chen CK. A comparison of Q-switched alexandrite laser and intense pulsed light for the treatment of freckles and lentigines in Asian persons: a randomized, physician-blinded, split-face comparative trial. J Am Acad Dermatol. 2006 May;54(5):804-10. doi: 10.1016/j.jaad.2006.01.012. PMID 16635661
- [Background] Kang HJ, Na JI, Lee JH, Roh MR, Ko JY, Chang SE. Postinflammatory hyperpigmentation associated with treatment of solar lentigines using a Q-Switched 532-nm Nd: YAG laser: a multicenter survey. J Dermatolog Treat. 2017 Aug;28(5):447-451. doi: 10.1080/09546634.2016.1254330. Epub 2016 Nov 15. PMID 27786580
- [Background] Hwang CY, Chen CC. Serial change in laser-induced optical breakdown by 1064-nm Nd:YAG picosecond laser. Photodermatol Photoimmunol Photomed. 2020 Jan;36(1):63-64. doi: 10.1111/phpp.12505. Epub 2019 Aug 29. No abstract available. PMID 31396986
- [Background] Wang YJ, Huang YK, Wang JY, Wu YH. In vivo characterization of large cell acanthoma by cellular resolution optical coherent tomography. Photodiagnosis Photodyn Ther. 2019 Jun;26:199-202. doi: 10.1016/j.pdpdt.2019.03.020. Epub 2019 Mar 30. No abstract available. PMID 30940575
- [Background] Farhi D, Falissard B, Dupuy A. Global assessment of psoriasis severity and change from photographs: a valid and consistent method. J Invest Dermatol. 2008 Sep;128(9):2198-203. doi: 10.1038/jid.2008.68. Epub 2008 Apr 17. PMID 18418412
- [Background] Arginelli F, Greco M, Ciardo S, Josse G, Rossi AB, Le Digabel J, Questel E, Chester J, Pellacani G. Efficacy of D-pigment dermocosmetic lightening product for solar lentigo lesions of the hand: A randomized controlled trial. PLoS One. 2019 May 1;14(5):e0214714. doi: 10.1371/journal.pone.0214714. eCollection 2019. PMID 31042723
- [Background] Pandya A, Berneburg M, Ortonne JP, Picardo M. Guidelines for clinical trials in melasma. Pigmentation Disorders Academy. Br J Dermatol. 2006 Dec;156 Suppl 1:21-8. doi: 10.1111/j.1365-2133.2006.07590.x. PMID 17176301
- [Background] van Geel N, Wolkerstorfer A, Ezzedine K, Pandya AG, Bekkenk M, Grine L, Van Belle S, Lommerts JE, Hamzavi I, Harris JE, Eleftheriadou V, Esmat S, Kang HY, Kumarasinghe P, Lan CE, Parsad D, Raboobee N, Flora Xiang L, Suzuki T, Prinsen CA, Taieb A, Picardo M, Speeckaert R; participants of the Rome International VGICC /VIS Workshop. Validation of a physician global assessment tool for vitiligo extent: Results of an international vitiligo expert meeting. Pigment Cell Melanoma Res. 2019 Sep;32(5):728-733. doi: 10.1111/pcmr.12784. Epub 2019 May 9. PMID 30945409